CLINICAL TRIAL: NCT02604836
Title: A Prospective, Open-Label, Multi-Center, Two-Part Study to Investigate Patient Satisfaction With Monthly Dosed Ibandronate Therapy in Women With Post-Menopausal Osteoporosis or Osteopenia Transitioned From Once-Weekly Alendronate or Risendronate
Brief Title: A Study of Ibandronate (Boniva) to Evaluate Satisfaction in Women With Post-Menopausal Osteoporosis or Osteopenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18056
Record Dates: First submitted 2015-11-06; First posted 2015-11-13 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Ibandronic Acid

ARMS (1):
- Ibandronate (Experimental): Participants will receive 150 milligrams (mg) of ibandronate as a film-coated tablet once-monthly.
  Interventions: Drug: Ibandronate

INTERVENTIONS:
Drug: Ibandronate — Film-coated oral ibandronate tablet (150 mg) once-monthly
  Other Names: Bonviva/Boniva

SUMMARY:
This study will investigate participant satisfaction (including compliance, preference, tolerability) with once-monthly Bonviva in women with post-menopausal osteoporosis or osteopenia transitioned from once-weekly alendronate or risedronate. The anticipated time on study treatment is 6 months, and the target sample size is 1776 individuals.

ELIGIBILITY:
Inclusion Criteria:

- Women who had been receiving once-weekly alendronate or risedronate for treatment or prevention of post-menopausal osteoporosis for greater than or equal to (>=) 3 months

Exclusion Criteria:

* Inability to stand or sit upright for >=60 minutes
* Hypersensitivity to bisphosphonates
* Inability to swallow a tablet whole
* Malignant disease diagnosed within previous 10 years (except resected basal cell cancer).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1711 (Actual)
Dates: Start 2004-06; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Part A: Number of participants who currently use weekly biphosphonate who answer "yes" to any of the questions in Candidate Identification Questionnaire (CIQ) | Up to 30 days prior to baseline visit
Part B: Number of participants who demonstrate improvement from their baseline satisfaction score after 6 months of ibandronate | 6 months
Part B: Percentage of participants who demonstrate improvement from their baseline satisfaction score after 6 months of ibandronate | 6 months

SECONDARY OUTCOMES:
Part B: Percentage of eligible weekly biphosphonate users at screening who elect to enter Part B | Screening visit
Part B: Percentage of participants who report an improved satisfaction score with monthly ibandronate compared to weekly alendronate or risendronate | 6 months
Part B: Percentage of participants who report preference to monthly ibandronate or weekly alendronate or risedronate | 6 months
Part B: Percentage of participants who have greater than or equal to (>=) 80 percent (%) compliance | 6 months
Part B: Percentage of participants who report an improvement in the gastrointestinal (GI) symptoms | 6 months
Part B: Percentage of participants by age and activity level who report high satisfaction according to Osteoporosis Patient Survey satisfaction Questionnaire (OPSAT-Q) | 6 months
Part B: Individual Domain scores from Osteoporosis Patient Survey satisfaction Questionnaire (OPSAT-Q) | Baseline and 6 months
Part B: Number of eligible weekly biphosphonate users at screening who elect to enter Part B | Screening Visit
Part B: Number of participants who report an improved satisfaction score with monthly ibandronate compared to weekly alendronate or risendronate | 6 months
Part B: Number of participants who report preference to monthly ibandronate or weekly alendronate or risedronate | 6 months
Part B: Number of participants who have >= 80% compliance | 6 months
Part B: Number of participants who report an improvement in the GI symptoms | 6 months
Part B: Number of participants by age and activity level who report high satisfaction according to Osteoporosis Patient Survey satisfaction Questionnaire (OPSAT-Q) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (131):
- United States (131):
  - Birmingham, Alabama
  - Columbiana, Alabama
  - Huntsville, Alabama
  - Mobile, Alabama
  - Montgomery, Alabama
  - Chandler, Arizona
  - Gilbert, Arizona
  - Paradise Valley, Arizona
  - Phoenix, Arizona
  - Tempe, Arizona
  - Tucson, Arizona
  - Carlisle, Arkansas
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Pine Bluff, Arkansas
  - Rogers, Arkansas
  - Searcy, Arkansas
  - Sherwood, Arkansas
  - Anaheim, California
  - Beverly Hills, California
  - Laguna Hills, California
  - Mission Viejo, California
  - Palm Desert, California
  - Palo Alto, California
  - Sacramento, California
  - San Diego, California
  - Tacoma, California
  - Vista, California
  - Westlake Village, California
  - Colorado Springs, Colorado
  - Lakewood, Colorado
  - Avon, Connecticut
  - Cromwell, Connecticut
  - Hamden, Connecticut
  - New London, Connecticut
  - Waterbury, Connecticut
  - Wilmington, Delaware
  - Aventura, Florida
  - Clearwater, Florida
  - DeLand, Florida
  - Fort Myers, Florida
  - Gainesville, Florida
  - Longwood, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Ocala, Florida
  - Palm Bay, Florida
  - Palm Harbor, Florida
  - Port Orange, Florida
  - Sarasota, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Decatur, Georgia
  - Rome, Georgia
  - Boise, Idaho
  - Coeur d'Alene, Idaho
  - Champaign, Illinois
  - Creve Coeur, Illinois
  - Peoria, Illinois
  - Evansville, Indiana
  - Arkansas City, Kansas
  - Newton, Kansas
  - Wichita, Kansas
  - Natchitoches, Louisiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Chelsea, Michigan
  - Detroit, Michigan
  - Saint Joseph, Michigan
  - Chaska, Minnesota
  - Jefferson City, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Billings, Montana
  - Omaha, Nebraska
  - Clifton, New Jersey
  - Middletown, New Jersey
  - New Brunswick, New Jersey
  - Princeton, New Jersey
  - Brooklyn, New York
  - East Syracuse, New York
  - New York, New York
  - Olean, New York
  - Rochester, New York
  - Stony Brook, New York
  - Durham, North Carolina
  - Fayetteville, North Carolina
  - Morehead City, North Carolina
  - Morganton, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Grand Forks, North Dakota
  - Beachwood, Ohio
  - Canfield, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Medford, Oregon
  - Portland, Oregon
  - Bala-Cynwyd, Pennsylvania
  - Langhorne, Pennsylvania
  - Philadelphia, Pennsylvania
  - Wyomissing, Pennsylvania
  - Charleston, South Carolina
  - Mt. Pleasant, South Carolina
  - Spartanburg, South Carolina
  - Bristol, Tennessee
  - Memphis, Tennessee
  - Murfreesboro, Tennessee
  - Nashville, Tennessee
  - Sevierville, Tennessee
  - Carrollton, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Denton, Texas
  - San Antonio, Texas
  - Wichita Falls, Texas
  - Norfolk, Virginia
  - Richmond, Virginia
  - Renton, Washington
  - Seattle, Washington
  - Spokane, Washington
  - Tacoma, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin